CLINICAL TRIAL: NCT05856578
Title: Nanjing Medical University, Nanjing First Hospital
Brief Title: Comparing the Efficacy of Mulberry Twig Alkaloid Tablet and Canagliflozin in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20220124-03
Record Dates: First submitted 2022-03-15; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Mulberry Twig (Ramulus Mori, Sangzhi) Alkaloid Tablet; Canagliflozin; Flash Glucose Monitoring （FGM）
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mulberry Twig Alkaloid Tablet (Experimental): Mulberry Twig (Ramulus Mori, Sangzhi) Alkaloid Tablet
  Interventions: Drug: Mulberry Twig Alkaloid Tablet
- Canagliflozin (Active Comparator): Canagliflozin
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Mulberry Twig Alkaloid Tablet — Mulberry Twig (Ramulus Mori, Sangzhi) Alkaloid Tablet 50mg po tid
  Other Names: Based on the original hypoglycemic treatment
  Arms: Mulberry Twig Alkaloid Tablet
Drug: Canagliflozin — Canagliflozin 100mg po qd
  Other Names: Based on the original hypoglycemic treatment
  Arms: Canagliflozin

SUMMARY:
The aim of the study is to investigate the efficacy and safety of Mulberry Twig (Ramulus Mori, Sangzhi) Alkaloid Tablet and Canagliflozin for 12 weeks in individuals with type 2 diabetes mellitus

DETAILED DESCRIPTION:
To compare the clinical efficacy, insulin resistance and blood glucose fluctuation of Mulberry Twig (Ramulus Mori, Sangzhi) Alkaloid Tablet and Canagliflozin in patients with type 2 diabetes mellitus using FGMS.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate and be able to sign informed consent prior to the trial.
* Patients with type 2 diabetes, aged 18-75 years old and BMI ≥18.0kg/m2.
* Treatment with one or two hypoglycemic drugs (in combination, the sulfonylureas dose should be less than half of the maximum dose).
* HbA1c : 7.0-9.0%.
* Subjects are able and willing to monitor peripheral blood sugar and regularity of diet and exercise.

Exclusion Criteria:

* Impaired liver and kidney function with ALT 2.5 times higher than the upper limit of normal value; Serum creatinine was 1.3 times higher than the upper limit of normal.
* Recurrent urinary tract infections.
* Drug abuse and alcohol dependence in the past 5 years.
* Patients with poor compliance and irregular diet and exercise.
* Systemic hormone therapy was used in the last three months.
* Patients with infection and stress within four weeks.
* Patients with pregnancy, lactation or pregnancy intention.
* Any other obvious conditions or associated diseases determined by the researcher: such as severe cardiopulmonary diseases, endocrine diseases, neurological diseases, tumors and other diseases, other pancreatic diseases, history of mental diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of FBG, PBG and HbA1c | 12 weeks
  The effects of Mulberry Twig Alkaloid Tablet and Canagliflozin on the concentration of FBG, PBG and HbA1c in patients with type 2 diabetes mellitus.
Concentration of MBG, TIR, TAR, TBR, MAGE, MBG and LAGE | 12 weeks
  The effects of Mulberry Twig Alkaloid Tablet and Canagliflozin on the changes of blood glucose fluctuations (including MBG, TIR, TAR, TBR, MAGE, MBG and LAGE) in patients with type 2 diabetes mellitus by FGM.

SECONDARY OUTCOMES:
Concentration of C-peptide, Insulin, glucagon and HOMA-IR | 12 weeks
  The effects of Mulberry Twig Alkaloid Tablet and Canagliflozin on C-peptide, Insulin, glucagon and HOMA-IR changes in patients with type 2 diabetes mellitus.
Concentration of the TC, TG, LDL, HDL and FFA | 12 weeks
  The effects of Mulberry Twig Alkaloid Tablet and Canagliflozin on concentration of blood lipid (including TC, TG, LDL, HDL, FFA) changes in patients with type 2 diabetes mellitus.
Concentration of adiponectin, leptin,IL-1,IL-6 andTNF-α | 12 weeks
  The effects of Mulberry Twig Alkaloid Tablet and Canagliflozin on the concentration of inflammatory factor(including adiponectin,leptin,IL-1,IL-6,TNF-α) changes in patients with type 2 diabetes mellitus.

OTHER OUTCOMES:
Fecal 16S rRNA gene sequencing | 12 weeks
  The effects of Mulberry Twig Alkaloid Tablet and Canagliflozin on types of intestinal flora changes in patients with type 2 diabetes mellitus by Fecal 16S rRNA gene sequencing.
Incidence of hypoglycemia | 12 weeks
  The effect of Mulberry Twig Alkaloid Tablet and Canagliflozin on the incidence of hypoglycemia in patients with type 2 diabetes mellitus by FGM.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, Study Director — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Jianhua Ma, Nanjing, China